CLINICAL TRIAL: NCT00644150
Title: Project Ai Shi Zi: Integrating HIV/STI Prevention and Treatment in China
Brief Title: Effectiveness of HIV/Sexually Transmitted Infection Training for Physicians in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas J. Coates, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH075639 (NIH); R01MH075639 (NIH); DAHBR 9A-ASG-P
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections; Gonorrhea; Chlamydia
Keywords: Risk Reduction Counseling; Anhui, China; HIV; STI
MeSH Terms: conditions — HIV Infections; Gonorrhea; Chlamydia Infections; Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Physicians of county level will receive Ai Shi Zi training provided by experts in the fields of HIV/STIs, behavioral counseling, and stigma reduction.
  Interventions: Behavioral: Physician Ai Shi Zi training
- 2 (Experimental): Physicians of township level will receive Ai Shi Zhi training provided by the county level physicians.
  Interventions: Behavioral: Physician Ai Shi Zi training
- 3 (Experimental): HIV/STI patients will receive standard of care and specialized care from physician participants trained in Ai Shi Zi.
  Interventions: Drug: Standard care; Behavioral: Patient risk-reduction counseling
- 4 (No Intervention): Physicians of county level who will not participate in Ai Shi Zi training
- 5 (No Intervention): Physicians of township level who will not participate in Ai Shi Zi training
- 6 (Sham Comparator): HIV/STI patients who will receive standard care only
  Interventions: Drug: Standard care

INTERVENTIONS:
Behavioral: Physician Ai Shi Zi training — This training uses a curriculum developed specifically for Project Ai Shi Zi and includes training in stigma; risk-reduction counseling; and quality HIV/STI diagnosis, treatment, and management. Physician training will consist of multiple components: an orientation workshop on fundamental knowledge and skills of HIV/STI treatment and prevention, a 3-month practice period, a 3-month post-practice seminar on preventive counseling, another 3-month practice period, and a 6-month post-practice seminar on clinical HIV and STI management. The practice periods will promote learning-by-doing to further enhance physicians' abilities to deliver high quality, integrated HIV/STI prevention and treatment. Post-practice seminars will allow participants to share experiences gained during the previous 3-month practice period.
  Arms: 1; 2
Drug: Standard care — If an STI is confirmed by a lab test, participants will receive standard of care treatment. Gonorrhea will be treated with a single dose of 250 mg of ceftriaxone sodium administered by intramuscular injection. If patients are allergic to ceftriaxone, they will be treated with azithromycin (2 g single oral dose). Chlamydia will be treated with azithromycin (1 g single oral dose).
  Arms: 3; 6
Behavioral: Patient risk-reduction counseling — On the initial visit, participants will receive HIV/STI risk-behavior counseling from the physician trained in Ai Shi Zi. The process is based on motivational interviewing techniques and will include discussing topics such as partner notification, HIV/STI prevention, and expected difficulties in changing behaviors. This risk-reduction model encourages the HIV/STI-infected or -uninfected person to develop a risk-reduction plan. The objective is to decrease the chance of infection for that individual and for others, too. Patients will develop a list of risk-reduction strategies to follow.
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of a physician training program, the Ai Shi Zi program, in improving HIV/sexually transmitted infection diagnosis, treatment, and management by Chinese physicians and in reducing the number of subsequent infections in their patients.

DETAILED DESCRIPTION:
HIV and sexually transmitted infections (STIs) are among the foremost public health concerns worldwide, with the number of infections continuing to rise significantly. Specifically, in China, the number of cases of HIV is estimated to rise from 650,000 in 2006 to more than 10 million by the year 2010. The reasons for the drastic increase may be associated with a lack of education about proper condom use and consequences of sexual risk behaviors and the existing stigma toward HIV/STI patients. Therefore, increased knowledge of HIV/STI prevention and treatment is necessary for both physicians and patients in China. A program that provides training in HIV/STI prevention, treatment, and management to physicians may be an effective means of enhancing their abilities to deliver high quality, integrated HIV/STI prevention and treatment. The Ai Shi Zi program, which provides training on stigma, risk-reduction counseling methods, and treatment skills to county and township level physicians in China, may be an effective means of implementing HIV/STI training. This study will evaluate the effectiveness of the Ai Shi Zi program in improving HIV/STI diagnosis, treatment, and management by Chinese physicians and in reducing the number of subsequent HIV/STI infections in their patients.

Participants in this study will include county level physicians and their patients and township level physicians. All physicians will first undergo baseline assessments that will include questions about knowledge of HIV/STI, capability of administering HIV/STI screening and risk-reduction counseling, and attitudes toward working with HIV/STI-infected individuals. Physicians will then be assigned randomly to receive the Ai Shi Zi program or no training.

Physician training in the Ai Shi Zi program will consist of multiple components: an orientation workshop on fundamental knowledge and skills of HIV/STI treatment and prevention, a 3-month practice period, a 3-month post-practice seminar on preventive counseling, another 3-month practice period, and a 6-month post-practice seminar on clinical HIV and STI management. Physicians will keep weekly journals during both 3-month practice periods, citing the most interesting or difficult STI or HIV case they experienced during the week. The practice periods will promote learning-by-doing to further enhance physicians' abilities to deliver high quality, integrated HIV/STI prevention and treatment. Both post-practice seminars will allow physicians to share experiences gained during the previous 3-month practice period. County level physicians will receive the seminar training from experts in the fields of HIV/STIs, behavioral counseling, and stigma reduction. After completing the first post-practice seminar, the county level physicians then, in turn, will present the training to the township level physicians. All physicians will undergo repeat baseline assessments at post-training; post-practice seminars; and Months 1, 2, and 15 after orientation.

Upon completion of the 6-month post-practice seminar, physicians will begin to implement the Ai Shi Zi program in their clinics. Each patient participant who seeks treatment from physician participants, who have received either Ai Shi Zi training or no training, will first undergo a test for chlamydia and gonorrhea. On this initial visit, the physicians who have received the Ai Shi Zi program will provide HIV/STI risk-behavior counseling to their patients. The counseling will include discussion of topics such as partner notification, HIV/STI prevention, expected difficulties in changing behaviors, and development of a risk-reduction plan. Patient participants will then return within 2 weeks to receive their test results and additional behavioral counseling. If the STI is confirmed by the lab test, patients will be treated with standard care and will be asked to complete an assessment. The assessment will include a 30-minute interview about HIV/STI-related knowledge, attitudes, beliefs, practices, service utilization, and risk behaviors. Nine months after baseline, patient participants will undergo a repeat interview.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

* Tests positive for the presence of gonorrhea or chlamydia
* Plans on living in current community for at least 9 months after study entry
* Willing to provide contact information for 9-month follow-up

Inclusion Criteria for County Level Physician Participants:

* Specializes in STI, obstetrics/gynecology, urology, infectious disease, or HIV care
* Minimum of 3 years of clinical experience as verified by practice supervisor
* Sees HIV/STI and related patients in his/her practice
* Willing to participate for the entire duration of the training, including secondary training stage

Inclusion Criteria for Township Level Physicians Participants:

* Minimum of 3 years of clinical experience as verified by practice supervisor
* Works in a high service volume area (among the top one-third within his/her host township health center)
* Sees HIV/STI and related patients in his/her practice
* Willing to participate for the entire duration of the training, including secondary training stage

Exclusion Criteria for All Participants:

* Presence of an obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation in the assessment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1373 (Actual)
Dates: Start 2007-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Scores from curriculum exams performed by physicians | Measured at Month 15

SECONDARY OUTCOMES:
Incidence of STIs in intervention patients | Measured at Month 9

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Coates, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Operario D, Wang D, Zaller ND, Yang MF, Blaney K, Cheng J, Hong Q, Zhang H, Chai J, Szekeres G, Galea J, Coates TJ. Effect of a knowledge-based and skills-based programme for physicians on risk of sexually transmitted reinfections among high-risk patients in China: a cluster randomised trial. Lancet Glob Health. 2016 Jan;4(1):e29-36. doi: 10.1016/S2214-109X(15)00249-1. PMID 26718807